CLINICAL TRIAL: NCT04222114
Title: A Two-stage,Multi-center,Open-label, Randomized,Controlled Trial Comparing the Efficacy and Safety of Intra-peritoneal Infusion of Catumaxomab and Treatment of Investigator Choice in Patients With Advanced Gastric Carcinoma With Peritoneal Metastasis
Brief Title: Comparing the Efficacy and Safety of Intra-peritoneal Infusion of Catumaxomab and Treatment of Investigator Choice in Patients With Advanced Gastric Carcinoma With Peritoneal Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LintonPharm Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0190415
Record Dates: First submitted 2020-01-05; First posted 2020-01-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Peritoneal metastasis; catumaxomab
MeSH Terms: conditions — Stomach Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catumaxomab group (Experimental)
  Interventions: Drug: Catumaxomab
- IC group (Active Comparator): IC group is defined as the localized supportive treatment which has been approved or recommended by local gastric cancer guidance to treat the peritoneal metastasis.
  Interventions: Drug: The treatment of investigator choice

INTERVENTIONS:
Drug: Catumaxomab — The starting dose of catumaxomab for intra-peritoneal infusion will be 10μg, gradually increased to 20μg, 50μg and 150μg, respectively. From the second cycle, catumaxomab will be changed to 20μg,50μg,150μg on days 1,4 and 8.
  Arms: Catumaxomab group
Drug: The treatment of investigator choice — the localized supportive treatment which has been approved or recommended by local gastric cancer guidance to treat the peritoneal metastasis.
  Arms: IC group

SUMMARY:
A total of 297 subjects are estimated to enroll in the study, with 15 eligible subjects enrolled in the 1st stage at most and 282 evaluable subjects in the 2nd stage. All subjects are adult patients with age over 18-year-old; they must be diagnosed with recurrent or metastatic gastric cancer with peritoneal metastasis at the time of enrollment; and failed at least prior two standard systemic anti-cancer therapies for recurrent or metastatic gastric cancer, before enrollment.

In the first stage, pharmacokinetic characteristics and preliminary safety of catumaxomab will be explored in Asian patients with gastric cancer ; in Cohort A, the enrolled subjects will receive the first infusion at 10μg on day 1, which will be increased to 20 μg, 50 μg and 150 μg on days 4, 8 and 11, respectively. 42 days are defined as a cycle. From the second cycle, catumaxomab will be changed to 20 μg, 50 μg, 150 μg on days 1, 4, 8 respectively. In Cohort B, 28 days are defined as a cycle. It is estimated to enroll 6 subjects in each cohort first.

In the second stage, approximate 282 subjects who meet the enrollment criteria are randomized into either catumaxomab infusion group (catumaxomab group) or treatment of investigator choice group (IC group), at a ratio of 2:1.

Subjects at the first and second stages will continue the treatment until one of the following conditions occurs:1)Significant progression of tumor lesions, including but not limited to peritoneal metastases lesions and/or ascites; 2)Intolerable toxicity; 3)The investigator believes that patients need to withdraw from the study and receive other treatment;4)death;5)Withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent forms have been provided.
2. Willing to be complaint with the study procedures during the study.
3. Male or female, age≥18years old when signing informed consents.
4. Histologically or cytologically confirmed as gastricadeno carcinoma.
5. Evaluable and/or non-evaluable lesions according to RECISTV1.1 criteria.
6. Diagnosed as gastric cancer with peritoneal metastases (Imaging finding, previous surgicalpathology, ascites/peritoneal effusion cytology positive).
7. Treatment failure after receiving at least prior two standard systemic anti-cancer therapies for recurrent or metastatic gastric cancer.
8. Recovered from any toxicity due to previous treatment (Grade 0-1 according to NCI-CTCAEv5.0).
9. Estimated survival length≥3months.
10. Eastern Oncology Cooperative Group(ECOG) performance status 0-2.
11. The laboratory test values during the screening period are in accordance with the following table：ANC(absolute neutrophil count)≥ 1.5 × 10^9/L， Hemoglobin≥ 80 g/L，Platelet≥ 100 × 10^9/L， Lymphocyte percentage≥13%，Serum Bilirubin≤ 1.25 x ULN(or 2.5 x ULN if there is Gilbert)， AST and ALT ≤ 2.5 × ULN without liver metastasis（or≤ 5 × ULN if liver metastasis ），Serum creatinine ≤ 2.0 mg/dL (or Calculated creatinine clearance≥30 mL/min).
12. For women of childbearing potential: use an efficient method for contraception at least 1 month prior to screening and agree to use this method for contraception during the study period and extended period specified after the study intervention.
13. For men with fertility potential: use condoms or other methods to ensure effective contraception for sexual partners.

Exclusion Criteria:

1. Known or suspected of being allergic to catumaxomab or similar antibodies.
2. Previously received anti-tumor treatments, including other anti-tumor investigational drugs, chemotherapy, immunotherapy, biological agents, hormone therapy, radiation therapy (except local radiation therapy for pain relief), etc., the interval between the last treatment and the first peritoneal infusion is ≤ 21days.
3. There is extensive liver metastasis(the tumor volume is estimated to be≥50% of the total liver volume by imaging).
4. Known tumor in tra-cranial metastases.
5. The following diseases have not been resolved to CTCAE grade 0-1 3 days before the first infusion:

   * Uncontrolled acute and chronic infections such as pneumonia, biliary infection, hepatitis B virus infection and hepatitis C virus infection,etc.;
   * Acute or chronic pancreatitis;
   * Diarrhea;
   * Dyspnea
6. NYHA Class 3 or 4.
7. Symptoms and signs of related cardiovascular diseases: including myocardial infarction, congestive heart failure,arrhythmia.
8. Known cerebrovascular accidents.
9. Intestinal obstruction occurred 30 days before the first dose.
10. Imaging diagnosis of portal vein obstruction, including tumor compression or portal thrombosis,cancer thrombus.
11. History of autoimmune diseases (e.g.,inflammatory bowel disease, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autologous hemolytic anemia, rheumatoid arthritis,etc.).
12. Patients with known HIV serology positive, hepatitis C infection and/or hepatitis B (Except the patients with HepBsAg or core antibody positive and responding to antiviral therapy against hepatitis B who are allowed to participate in the study; Notes: HepBsAg-negative patients at screening, or patients are undergoing treatment with interferon-2a [IFN] or peginterferon-2a [Peg-IFN] and hepatitis B virus [HBV] DNA < 2000 international units [IU], or subjects who are receiving nucleoside [acid] analogues at screening and HBV DNA below the lower limit of normal [LLN] are eligible to participate in the study).
13. Pregnancy or breast feeding during study treatment and follow-up.
14. Patients with confirmed history of neurological or psychotic disorders, including epilepsy or dementia.
15. Other serious systemic conditions that may limit the patient's participation in this study (eg uncontrolled diabetes, cardiovascular and cerebrovascular disease, severe gastrointestinal disease,etc.).
16. Any other condition that, in the discretion of the investigator will make patients exposed to unnecessary risks and unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 1 year
  Defined as the time from randomization to death for anyreason.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year
  According to RECIST V1.1 criteria, defined as the timefrom randomization to progression disease (PD) or death for any reason,which ever occurs first.
Progression free interval of peritoneal metastatic lesions | 1 year
  to subjects with ≥300 ml of ascites, defined as the time from first intra-peritoneal infusion to ascites progression based on the five--point method2; to subjects without ascites or <300 ml, it is defined as the time from the first intra-peritoneal infusion to thetimeof progression oftheintra-peritoneal lesion according to theRECISTV1.1 criteria.
Objective Response Rate (ORR) | 1 year
  According to RECIST V1.1 criteria, defined as the proportion of subjects with response achieving CR or PR;
Clinical Benefit Rate(CBR) | 1 year
  According to RECIST V1.1 criteria,defined as the proportion of subjects with response achieving SD,PR or CR;
Duration of Response (DoR) | 1 year
  According to RECIST V1.1 criteria, defined as the time from the response to the confirmation of PD
Ascites Remission Duration | 1 year
  Defined as the time from the 1st as cites remission to as cites progression,according to the five-point method.
The incidence and severity of treatment-emergent adverse events (TEAEs) in the catumaxomab and IC groups | 1 year
  Compared according to the National Cancer Institute Common Terminology Standard for Adverse Events (NCI-CTCAE)v5.0.
Incidence of DLT | 1 year
  it will be evaluated in the first stage only. It is defined as the incidence of DLT from the first infusion to 6 weeks after wards.
The incidence of anti-drug antibodies(ADA) to catumaxomab in serum | 1 year
  The incidence of anti-drug antibodies(ADA) to catumaxomab in serum
Tendency of theperipheral blood lymphocyte counts change associated with the intra-peritoneal infusion of catumaxomab | 1 year
  Tendency of theperipheral blood lymphocyte counts change associated with the intra-peritoneal infusion of catumaxomab

CONTACTS AND LOCATIONS:
Locations (13):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Bethune Hospital of Jilin University., Jilin, Jilin
- South Korea (4):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Cheng Kung University Hospital, Tainan